CLINICAL TRIAL: NCT02828917
Title: Multi-center Study for Evaluating the Safety and Efficacy of the MedJ-01 Ridaforolimus Eluting Coronary Stent System (MedJ-01) In Coronary Stenosis Trial
Brief Title: MedJ-01 Ridaforolimus Eluting Coronary Stent System Trial (JNIR)
Acronym: JNIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medinol Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JNIR01
Record Dates: First submitted 2016-07-03; First posted 2016-07-12 (Estimated); Results first posted 2020-09-24 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: de Novo or Restenosis Lesions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MedJ-01 drug eluting stent (Experimental): MedJ-01 Ridaforolimus eluting coronary stent system
  Interventions: Device: MedJ-01 Ridaforolimus Eluting Coronary Stent System

INTERVENTIONS:
Device: MedJ-01 Ridaforolimus Eluting Coronary Stent System

SUMMARY:
MedJ-01 Ridaforolimus Eluting Coronary Stent System is a single use device/drug combination product comprising:

* A mounted Cobalt Chromium (CoCr) alloy based stent
* A Rapid Exchange (RX) Coronary System Delivery System
* A Poly n-butyl methacrylate (PBMA) and CarboSil®Polymer matrix coating
* Ridaforolimus drug - CAS Registry Number: 572924-54-0 MedJ-01 is indicated for improving coronary luminal diameter in patients with symptomatic heart disease due to lesions in vessels with reference diameters of 2.5 mm to 4.25 mm, including complex lesions.

JNIR01 is aimed at assessing TLF at one year with the MedJ-01 stent in a Japanese patient population to show equivalence to the results of the BIONICS Trial.

DETAILED DESCRIPTION:
This study aims to evaluate MedJ-01 safety and efficacy for de novo or restenosis lesion with target vessel diameter of 2.5mm to 4.25, for subjects undergoing coronary artery stent implantation. The target population is subjects undergoing PCI for angina (stable or unstable), silent ischemia (in absence of symptoms a visually estimated target lesion diameter stenosis of ≥70%, a positive non-invasive stress test, or FFR ≤0.80 must be present), NSTEMI, and recent subacute STEMI (>72 hours from initial presentation and stable). Complex lesions are allowed. A maximum of two target vessels and two lesions per vessel may be treated (two lesions separated by up to 10 mm that can be covered by a single stent are considered as one lesion); the total planned study stenting in the coronary tree cannot exceed 100 mm.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with indication for PCI including angina (stable/unstable), silent ischemia (in absence of symptoms a visually estimated target lesion diameter stenosis of ≥70%, a positive non-invasive stress test, or FFR ≤0.80 must be present), NSTEMI, or recent subacute STEMI. For subacute STEMI the time of presentation to the first treating hospital, whether a transfer facility or the study hospital, must be >72 hours prior to enrollment and enzyme levels (CK-MB or Troponin) demonstrating that either or both enzyme levels have peaked.
2. Non-target vessel PCI are allowed prior to enrollment depending on the time interval and conditions as follows:

   * During Baseline Procedure:

     * PCI of non-target vessels performed during the baseline procedure itself immediately prior to enrollment if successful and uncomplicated defined as: <50% visually estimated residual diameter stenosis, TIMI Grade 3 flow, no dissection ≥ NHLBI type C, no perforation, no persistent ST segment changes, no prolonged chest pain, no TIMI major or BARC type 3 bleeding.
     * Less than 24 hours prior to Baseline Procedure:
   * Not allowed (see exclusion criterion #2).

     * 24 hours-30 days prior to Baseline Procedure:
     * PCI of non-target vessels 24 hours to 30 days prior to enrollment if successful and uncomplicated as defined above.
   * In addition, in cases where non-target vessel PCI has occurred 24-72 hours prior to the baseline procedure, at least 2 sets of cardiac biomarkers must be drawn at least 6 and 12 hours after the non-target vessel PCI.
   * If cardiac biomarkers are initially elevated above the local laboratory upper limit of normal, serial measurements must demonstrate that the biomarkers are falling.

     * Over 30 days prior to Baseline Procedure:
     * PCI of non-target vessels performed greater than 30 days prior to procedure whether or not successful and uncomplicated.
3. Patient is willing and able to provide informed written consent and comply with follow-up visits and testing schedule.

   Angiographic inclusion criteria (visual estimate):
4. Target lesion(s) must be located in a native coronary artery with visually estimated diameter of ≥2.5 mm to ≤4.25 mm.
5. Complex lesions are allowed including calcified lesions (lesion preparation with scoring/cutting and rotational atherectomy are allowed), presence of thrombus that is non-occlusive and does not require thrombectomy, CTO, bifurcationlesions (except planned dual stent implantation), ostial RCA lesions, tortuous lesions, bare metal stent restenotic lesions, protected left main lesions.
6. Overlapping stents are allowed with the investigational device (MedJ-01).

Exclusion Criteria:

1. STEMI within 72 hours (subacute) of initial time of presentation to the first treating hospital, whether at a transfer facility or the study hospital or in whom enzyme levels (either CK-MB or Troponin) have not peaked.
2. PCI within the 24 hours preceding the baseline procedure.
3. Non-target lesion PCI in the target vessel within 12 months of the baseline procedure.
4. History of stent thrombosis.
5. Cardiogenic shock (defined as persistent hypotension (systolic blood pressure <90 mm/Hg for more than 30 minutes) or requiring pressors or hemodynamic support, including IABP.
6. Subject is intubated.
7. Known LVEF <30%.
8. Relative or absolute contraindication to DAPT for 12 months (including planned surgeries that cannot be delayed)
9. Subject has an indication for chronic oral anticoagulant treatment (with either vitamin K antagonists or novel anticoagulants - NOACs)
10. Calculated creatinine clearance <30 mL/min using Cockcroft-Gault equation.
11. Hemoglobin <10 g/dL.
12. Platelet count <100,000 cells/mm3 or >700,000 cells/mm3.
13. White blood cell (WBC) count <3,000 cells/mm3.
14. Clinically significant liver disease.
15. Active peptic ulcer or active bleeding from any site.
16. Bleeding from any site within the prior 8 weeks requiring active medical or surgical attention.
17. If femoral access is planned, significant peripheral arterial disease which precludes safe insertion of a 6F sheath.
18. History of bleeding diathesis or coagulopathy or will refuse blood transfusions.
19. Cerebrovascular accident or transient ischemic attack within the past 6 months, or any permanent neurologic defect attributed to CVA.
20. Known allergy to the study stent components e.g. cobalt, nickel, chromium, Carbosil®, PBMA, or limus drugs (ridaforolimus, zotarolimus, tacrolimus, sirolimus, everolimus, or similar drugs or any other analogue or derivative or similar compounds).
21. Known allergy to protocol-required concomitant medications such as aspirin, or DAPT (Drugs that inhibit P2Y12 such as clopidogrel and prasugrel), or heparin, or iodinated contrast that cannot be adequately pre-medicated.
22. Any co-morbid condition that may cause non-compliance with the protocol (e.g. dementia, substance abuse, etc.) or reduced life expectancy to <24 months (e.g. cancer, severe heart failure, severe lung disease).
23. Patient is participating in any other investigational drug or device clinical trial that has not reached its primary endpoint, or plans to participate in any clinical trial.
24. Women who are pregnant or breastfeeding (women of child-bearing potential, defined as females of childbearing potential if they have not undergone a permanent contraceptive operation or they are not postmenopausal, must have a negative pregnancy test within one week before treatment. Permanent contraceptive operation is defined as: hysterectomy, hysterosalpingectomy, or bilateral oophorectomy. The status of a female should be considered as postmenopausal when she has not had a period for 12 consecutive months without an alternative medical cause).
25. Women who intend to become pregnant within 12 months after the baseline procedure (women of child-bearing potential who are sexually active must agree to use a reliable method of contraception from the time of screening through 12 months after the baseline procedure).
26. Patient has received an organ transplant or is on a waiting list for an organ transplant.
27. Patient is receiving or scheduled to receive chemotherapy within 30 days before or any time after the baseline procedure.
28. Patient is receiving oral or intravenous immunosuppressive therapy or has known life-limiting immunosuppressive or autoimmune disease (e.g., HIV). Corticosteroids are allowed.

    Angiographic Exclusion Criteria (visual estimate):
29. Target lesions in more than two (2) major coronary arteries (i.e., two of LAD, LCX, RCA) and their respective branches (the Ramus Intermedius is defined as a branch of the LCX).
30. More than two target lesions per target vessel are planned (two lesions separated by less than 10 mm that can be covered by a single stent are considered as one lesion).
31. More than 100 mm length of planned study stenting in the entire coronary tree.
32. Occlusive thrombus and/or a thrombus requiring thrombectomy in a target vessel.
33. Unprotected left main lesions ≥30%, or planned unprotected left main intervention.
34. Ostial LAD or LCX lesions (stenting of any diseased segment within 5 mm of the unprotected left main coronary artery).
35. Bifurcation lesions with planned dual stent implantation.
36. Stenting of lesions due to DES restenosis.
37. Another lesion in a target or non-target vessel (including all side branches) is present that requires or has a high probability of requiring PCI within 12 months after the baseline procedure.
38. Target lesion exists in bypass graft vessels.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2017-01-16 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2022-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shigeru Saito, MD, Principal Investigator — Shonan Kamakura General Hospital; Seiji Yamazaki, MD, Principal Investigator — Sapporo Higashi Tokushukai Hospital; Atsuo Namiki, MD, Principal Investigator — Kanto Rosai Hospital; Yoshisato Shibata, MD, Principal Investigator — Miyazaki Medical Association Hospital; Satoru Otsuji, MD, Principal Investigator — Higashi Takarazuka Satoh Hospital; Shigeu Nakamura, MD, Principal Investigator — Kyoto Katsura Hospital; Akihiko Takahashi, MD, Principal Investigator — Takahashi Hospital; Tomohiro Kawasaki, MD, Principal Investigator — Shin Koga Hospital; Yasuhiro Makita, MD, Principal Investigator — Hospital Hakodate Hokkaido; Takeshi Serikawa, MD, Principal Investigator — Saiseikai Fukuoka General Hospital
Locations (1):
- Shonan Kamakura General, Kamakura, Kanagawa, Japan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MedJ-01 Drug Eluting Stent
Started | 104
Completed | 104
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | MedJ-01 Drug Eluting Stent
Number analyzed (Participants) | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 77
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 83
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 104
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 104
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 104

OUTCOME MEASURES:

1. Primary Outcome: Target Lesion Failure (TLF)
Description: TLF is defined as the composite of cardiac death, target vessel-related myocardial infarction, or ischemia-driven target lesion revascularization.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | MedJ-01 Drug Eluting Stent
Number analyzed (Participants) | 104
Participants | 2

2. Secondary Outcome: Device Success at Time of Baseline Procedure
Description: Device Success at time of baseline procedure- outcome
Time Frame: 30 days, 6 months, and 1, 2, 3, 4 and 5 years
Reporting Status: Not Posted

3. Secondary Outcome: Lesion Success at Time of Baseline Procedure
Description: Lesion Success at time of baseline procedure- outcome
Time Frame: 30 days, 6 months, and 1, 2, 3, 4 and 5 years
Reporting Status: Not Posted

4. Secondary Outcome: Procedure Success at Time of Baseline Procedure
Description: Procedure Success at time of baseline procedure- outcome
Time Frame: 30 days, 6 months, and 1, 2, 3, 4 and 5 years
Reporting Status: Not Posted

5. Secondary Outcome: TLF
Description: TLF- target lesion failure
Time Frame: 30 days, 6 months, and 2, 3, 4 and 5 years
Reporting Status: Not Posted

6. Secondary Outcome: Major Adverse Cardiac Events (MACE)
Description: MACE is the composite rate of cardiac death, any MI or ischemia-driven TLR
Time Frame: 30 days, 6 months, and 1, 2, 3, 4 and 5 years
Reporting Status: Not Posted

7. Secondary Outcome: Target Vessel Failure (TVF)
Description: the composite rate of death, target vessel related MI or ischemia-driven TVR
Time Frame: 30 days, 6 months, and 1, 2, 3, 4 and 5 years
Reporting Status: Not Posted

8. Secondary Outcome: All-cause Mortality
Description: All-cause mortality outcome
Time Frame: 30 days, 6 months, and 1, 2, 3, 4 and 5 years
Reporting Status: Not Posted

9. Secondary Outcome: Cardiac Death
Description: Cardiac Death outcome
Time Frame: 30 days, 6 months, and 1, 2, 3, 4 and 5 years
Reporting Status: Not Posted

10. Secondary Outcome: Myocardial Infarction
Description: Myocardial Infarction (MI)
Time Frame: 30 days, 6 months, and 1, 2, 3, 4 and 5 years
Reporting Status: Not Posted

11. Secondary Outcome: Target Vessel Related MI
Description: Target Vessel Related MI outcome
Time Frame: 30 days, 6 months, and 1, 2, 3, 4 and 5 years
Reporting Status: Not Posted

12. Secondary Outcome: Ischemia-driven TLR
Description: Ischemia-driven TLR outcome
Time Frame: 30 days, 6 months, and 1, 2, 3, 4 and 5 years
Reporting Status: Not Posted

13. Secondary Outcome: Ischemia-driven TVR
Description: Ischemia-driven TVR outcome
Time Frame: 30 days, 6 months, and 1, 2, 3, 4 and 5 years
Reporting Status: Not Posted

14. Secondary Outcome: Stent Thrombosis
Description: ARC definite and probable
Time Frame: 30 days, 6 months, and 1, 2, 3, 4 and 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The Investigator monitored the occurrence of adverse events or device deficiencies for each subject during the whole course of the trial, visits: baseline and post procedure, 30 days, 6 months, 1 year, 2 years, 3 years, 4 years and 5 years.
Arm/Group | MedJ-01 Drug Eluting Stent
All-Cause Mortality (participants affected / at risk) | 1/104
Serious Adverse Events (participants affected / at risk) | 21/104
Other Adverse Events (participants affected / at risk) | 59/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MedJ-01 Drug Eluting Stent (N=104)
cardiac disorders (Cardiac disorders) | 7 (7)
Eye disorders (Eye disorders) | 2 (2)
Gastrointestinal disorders (Gastrointestinal disorders) | 7 (8)
General disorders and administration site conditions (General disorders) | 3 (3)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 2 (2)
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Renal and urinary disorders (Renal and urinary disorders) | 1 (1)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 (1)
Vascular disorders (Vascular disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MedJ-01 Drug Eluting Stent (N=104)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 2 (2)
Cardiac Disorders (Cardiac disorders) | 15 (15)
Eye disorders (Eye disorders) | 3 (4)
Gastrointestinal disorders (Gastrointestinal disorders) | 14 (20)
General disorders and administration site conditions (General disorders) | 12 (14)
Hepatobiliary disorders (Hepatobiliary disorders) | 1 (1)
Infections and infestations (Infections and infestations) | 17 (20)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 11 (13)
Investigations (Investigations) | 2 (2)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 2 (2)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 5 (5)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (5)
Nervous system disorders (Nervous system disorders) | 8 (8)
Psychiatric disorders (Psychiatric disorders) | 1 (1)
Renal and urinary disorders (Renal and urinary disorders) | 3 (4)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 12 (12)
Vascular disorders (Vascular disorders) | 5 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-09-18): https://cdn.clinicaltrials.gov/large-docs/17/NCT02828917/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/17/NCT02828917/SAP_001.pdf